CLINICAL TRIAL: NCT06315036
Title: Effects of Developmental Gymnastics Exercise Program on Preschoolers' Motor Skills: a Randomized Controlled Trial
Brief Title: Effects of Developmental Gymnastics on Preschoolers' Motor Skills
Acronym: GymKids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Dragan Marinkovic, Lead Investigator, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32/2021
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Motor Activity; Child Development; Exercise
Keywords: Gymnastics; Kindergarten; Sports school; TGMD-2
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Developmental gymnastics (DG) (Experimental): Developmental gymnastics group of participants
  Interventions: Other: Developmental gymnastics
- Control (CG) (No Intervention): Control group of participants

INTERVENTIONS:
Other: Developmental gymnastics — The DG exercise program ran from September 15, 2021, to May 15, 2022, in a well-equipped gymnasium. Led by trained teachers and gymnastics experts, sessions were held twice weekly (Tuesday and Thursday) for 60 minutes. The program focused on stability, locomotor skills, and manipulation, introducing children to DG fundamentals. It included circuit and station training, obstacle courses, and gradually increased exercise complexity. Sessions comprised a 15-minute warm-up, a 40-minute main session with skill practice and conditioning, and a 5-minute cool-down. The atmosphere was positive and friendly, with kid-friendly music and adapted procedures from previous research.
  Arms: Developmental gymnastics (DG)

SUMMARY:
Background: During childhood, physical activity (PA) is considered indispensable for developing motor skills through movement in the early stages of human development. Being active helps individuals develop fine and gross motor skills (GMS) by promoting an active lifestyle. Notably, this phase, characterized by regular PA and attaining motor competence, is associated with many health-related benefits. Early motor intervention programs have garnered attention for their positive influence on children's motor skills, as evidenced by various studies. A spectrum of more specialized methods is available alongside these general approaches, including programs designed to augment the time dedicated to general PA within school environments. Previous research has demonstrated the efficacy of incorporating experimental exercise interventions, grounded in enjoyable activities and game drills, into the curriculum, significantly improving children's basic motor skills. Many research articles have explored the impact of developmental gymnastics (DG) on children's fitness, indicating that gymnastics training can produce numerous beneficial outcomes for children's physical fitness.

Method and Materials: Three hundred preschool children were assigned to either a gender-balanced group participating in a DG exercise program (EG; n=99) or a control group (CG; n=121). While individuals in the CG followed three structured extracurricular physical activities per week in kindergarten, the EG participants received 60 minutes of the DG exercise program two days a week. The Test of Gross Motor Development-2 (TGMD-2) was used to assess GMS.

Aim: The study aimed to determine if participation in a structured DG program could improve GMS among preschool children compared to those in a group that attended extracurricular physical activities in a kindergarten.

DETAILED DESCRIPTION:
Study design Developmental gymnastics (DG) presents a specialized form of gymnastics focusing on individuals' physical, cognitive, and motor development, typically children. The study aimed to determine the effects of DG, which lasts nine months, on preschoolers' gross motor skills (GMS). The study presents an Interventional study to improve motor abilities, and the main objective is prevention. The study model is parallel with two groups.

Participants The initial sample of respondents (n=350) was recruited through an open project application lasting two months (from 1 July 2021 to 1 September 2021), from which 300 preschool children aged 4-7 were selected for this randomized, controlled interventional study. The recruitment process was completed after the selection process, and the optimal sample of subjects was filled out. The study sample underwent stratified randomization, resulting in the division into either EG (Experimental Group - 1) or CG (Control Group - 2). When stratifying, researchers used proportionate sampling to maintain the correct proportions of genders in every group. The intervention program started with a group of 150 children in EG, and at the same time, 150 children in CG started a kindergarten educational program in a Preschool Institution. Throughout the nine months of the experimental program, 51 children from the intervention group and 29 from the control group were excluded from the final analyses due to injury, flu, illness, or attendance at classes falling below 80%. Finally, 99 children (54 boys & 45 girls) who composed the EG and 121 children (64 boys & 57 girls) who composed the CG were analyzed for the effects of the DG. After nine months, a total of 220 participants were included in the final analysis. The parents or guardians of each child provided written informed consent, and the study received approval from the institutional ethics committee at the Faculty of Sport and Physical Education, University of Novi Sad (ethical approval number: 46-06-04/2020-1).

Testing procedures

Secondary outcome - Anthropometric measures Anthropometric data, including height and weight, were collected before the motor competence and physical fitness assessment. Following Martin's guidelines, body height was measured using a fixed anthropometer (GPM Anthropometer 100; DKSH Switzerland Ltd., Zurich, Switzerland; ± 0.1 cm). Body mass was measured with a digital balance (BC1000, Tanita, Japan; ± 0.1 kg), following the guidelines proposed by the International Biological Program (IBP). The body mass index (BMI) was calculated using the weight/height^2 (kg/m^2) formula based on the provided height and weight values.

Primary outcome - TGMD-2 The Test of Gross Motor Development - 2 (TGMD-2) is a standardized test to assess gross motor functioning in children aged 3 through 10. Researchers have previously utilized the TGMD-2, which demonstrates high reliability and minimal test error, instilling confidence in its application. The TGMD-2 measures 12 fundamental motor skills divided into two subcategories. The locomotor subtest consists of six skills: run, hop, gallop, leap, horizontal jump, and slide. The object control subtest includes six skills: hitting a stationary ball, dribbling while stationary, catching, kicking, throwing overhand, and rolling underhand. Motor competence was assessed with the TGMD-2 using the detailed instruction manual by examiners trained in physical education with prior experience in TGMD-2 measurements. Experienced researchers in test assessments coordinated and supervised the assessments. Each test took approximately 15-20 minutes and was performed indoors. The assessments were carried out, recorded, and coded at the Gymnastics Center, Faculty of Sport and Physical Education, University of Novi Sad, Serbia, from 1. September 2021 to 15. September 2021. Following a visual demonstration, each participant performed all 12 skills of the TGMD-2, receiving one practice attempt and two assessment trials for each skill. Each skill consists of three to five performance criteria, with one score assigned if the criterion is present and zero if not. Total scores for each skill and subtest were calculated, ranging from 0 to 48.

Interventions The Developmental Gymnastics Exercise Program The nine-month DG exercise program (from 15 September 2021 to 15 May 2022) was conducted indoors in a well-equipped gymnasium. Trained physical education teachers and gymnastics experts led the training sessions twice weekly (on Tuesday and Thursday) without a break throughout the experimental period. Each session lasted for 60 minutes and covered a range of gymnastics activities and exercises, with each week focusing on specific categories of GMS, such as stability (trunk strength), locomotor skills (running, hopping, skipping), and manipulation (ball skills). The program also introduced children to fundamental elements of DG and was meticulously structured, incorporating frontal and group work, primarily circuit training (polygon) or repetitive (station) training. Obstacle courses were designed to incorporate various gymnastic apparatus and props, encouraging problem-solving through gymnastic and athletic exercises and elementary games. The number of repetitions, sets, and complexity of exercises and routines gradually increased in the central part of the session as children could perform them quickly, accompanied by external cues such as sweating, blushing, spontaneous breaks, and heart rates. The training structure consisted of three parts: I) A 15-minute warm-up with diverse movements, speed-varied exercises, activities for flat feet, stretching, corrective and preventive exercises for posture improvement, and a focus on proper performance awareness. II) The central part lasted 40 minutes and included reviewing and practicing previous skills, introducing and practicing new skills, engaging in competitive activities, and conditioning exercises. III) A 5-minute cool-down involving stretching, coaching feedback, and informal discussion about sports, exercise, and daily activities. A positive and friendly atmosphere was maintained throughout each training session, accompanied by suitable kids' music, especially during the introduction and preparation phases. Basic principles and procedures were adapted from previous research.

In contrast, the CG adhered to their routine, engaging in three structured extracurricular physical activity sessions per week, each lasting approximately 45 minutes. A physical education specialist and a kindergarten teacher led these sessions. They were designed to enhance fundamental locomotor skills (e.g., hopping, skipping, jumping, crawling, and navigating obstacles) and manipulative skills involving balls, bricks, and toys. The primary objective was to create an environment where children could enjoy and have fun during exercise. According to the National Program for Kindergarten Physical Education Classes, the standardized program predominantly featured frontal and group activities, encompassing traditional games and dances, and included different training forms. The authors did not thoroughly provide detailed information about the intervention program.

Statistical analyses Unless otherwise specified, data are presented as mean and 95% confidence intervals [95% CIs]. An independent samples t-test was conducted to examine whether the baseline study outcomes varied among the groups. Normality was confirmed using the Kolmogorov-Smirnov test, and homogeneity of variances and covariance matrices were accepted through Levene's and Box's tests, respectively. The raw scores of each study outcome were modeled using a 2x (girls vs. boys), 2x (EG vs. CG), and 2 (initial vs. final testing) mixed ANCOVA (Model 1) to test confounding effects of gender, age, and BMI on intervention effects. The main effects of gender, age, and BMI were inspected to assess whether the study outcomes depended on these factors. This examination aimed to determine whether gender, age, and BMI could control the effects of the DG program on the study outcomes. Hence, respecting the significance of control variables effects (p≤0.05), each study outcome was modeled using either a 2x (girls vs. boys) 2x (EG vs. CG) 2 (initial vs. final testing) mixed ANCOVA with age and BMI or only with age to find whether study outcome mean changes [95% CIs] from initial to final testing depended on whether subjects completed DG program or not (Model 2). Potential gender confounding effects on changes in the study outcomes were assessed by examining a time*group*gender interaction effect, followed by a time*group interaction effect for boys and girls, respectively. The time*group interaction effects allowed the evaluation of DG program effects followed by the simple main effects of time, which designated mean changes [95% CIs] from initial to final testing for each group. In addition, the parameters (beta coefficients, β and partial eta2, ŋ2) of ANCOVA models were estimated. Games-Howel tests corrected multiple comparisons, and a p-value of ≤0.05 designated statistical significance. Partial eta squared (partial ŋ2) is reported as a measure of effect size and classified as small (0.01), medium (0.06), and large (0.14), according to Cohen. All analyses were conducted using SPSS (v.23, IBM Corporation, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

* No injuries within the past six months
* No other medical conditions, including COVID-19
* No scheduled physical activity in the previous three months
* Considered valid for the experimental programs if participants completed at least 80% of all training sessions.

Exclusion Criteria:

* History of neurological or musculoskeletal disorders
* Clinical conditions that could affect balance, such as motor disorders, diabetes, heart disease, stroke, vision problems, thyroid issues, or issues with nerves or blood vessels.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Test of gross motor development (tgmd-2): Locomotor Skills - Run | Nine months
  EQUIPMENT/CONDITIONS: A minimum of 50 feet of clear space and masking tape, chalk, or other marking device.
  DIRECTIONS: Mark off two lines 50 feet apart. Instruct student to "run fast" from one line to the other.
  PERFORMANCE CRITERIA:
  Brief period where both feet are off the ground! Arms in opposition to legs, elbows bent. Foot placement near or on line (not flat footed) Non-support leg bent approximately 90 degrees (close to buttocks).
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Locomotor skills - Gallop | Nine months
  EQUIPMENT/CONDITIONS: A minimum of 30 feet of clear space. DIRECTIONS: Mark off two lines 30 feet apart. Tell student to gallop from one line to the other three times. Tell student to gallop leading with one foot and then the other.
  PERFORMANCE CRITERIA:
  A step forward with the lead foot followed by a step with the trailing foot to a position adjacent to or behind the led foot.
  Brief period where both feet are off the ground. Arms bent and lifted to waist level. Able to lead with right and left foot.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Locomotor skills - Hop | Nine months
  EQUIPMENT/CONDITIONS: A minimum of 15 feet of clear space. DIRECTIONS: Ask the student to hop three times, first on one foot and then on the other.
  PERFORMANCE CRITERIA:
  Foot of non-support leg is bent and carried in back of the body. Non-support leg swings in pendular fashion to produce force. Arms bent at elbows and swing forward on take-off. Able to hop on the right and left foot.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Locomotor skills - Leap | Nine months
  EQUIPMENT/CONDITIONS: A minimum of 30 feet of clear space. DIRECTIONS: Ask the student to leap. Tell the student to take large steps by leaping from one foot to the other.
  PERFORMANCE CRITERIA:
  Take off on one foot and land on the opposite foot. A period where both feet are off the ground (longer than running). Forward reach with arm opposite the lead foot.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Locomotor skills - Horizontal jump | Nine months
  * EQUIPMENT/CONDITIONS:** A minimum of 10 feet of clear space and masking tape or another marking device.
  * DIRECTIONS:** Mark off a starting line on the floor, mat, or carpet. Have the student start behind the line. Instruct the student to "jump far."
  **PERFORMANCE CRITERIA:**
  1. Preparatory movement includes flexion of both knees with arms extended behind the body.
  2. Arms extend forcefully forward and upward, reaching full extension above the head.
  3. Take off and land on both feet simultaneously.
  4. Arms are brought downward during landing.
  **EXPERT SCORING:**
  1. Require three trials.
  2. Observe and focus on performance criteria.
  3. Score "1" for correct performance on two out of three trials, otherwise score "0."
Test of gross motor development (tgmd-2): Locomotor skills - skip | Nine months
  EQUIPMENT/CONDITIONS: A minimum of 30 feet of clear space and masking tape, or other marking device.
  DIRECTIONS: Mark off two lines 30 feet apart. Tell the student to skip from one line to the other three times.
  PERFORMANCE CRITERIA:
  A rhythmical repetition of the step-hop on alternate feet. Foot of non-support leg carried near surface during hop phase. Arms alternately moving in opposition to legs at about waist level.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Locomotor skills - slide | Nine months
  * EQUIPMENT/CONDITIONS:** A minimum of 30 feet of clear space and masking tape or another marking device.
  * DIRECTIONS:** Mark off two lines 30 feet apart. Instruct the student to slide from one line to the other three times, facing the same direction.
  **PERFORMANCE CRITERIA:**
  1. Body turned sideways to the desired direction of travel.
  2. A step sideways followed by a slide of the trailing foot next to the lead foot.
  3. A short period where both feet are off the floor.
  4. Able to slide to the right and left sides.
  **EXPERT SCORING:**
  1. Require three trials.
  2. Observe and focus on performance criteria.
  3. Score "1" for correct performance on two out of three trials, otherwise score "0."
Test of gross motor development (tgmd-2): Object control skill- two-hand strike | Nine months
  EQUIPMENT/CONDITIONS: A 4-6-inch light-weight ball and plastic bat. DIRECTIONS: Toss the ball softly to the student at about waist level. Tell the student to hit the ball "hard." Count only those tosses that are between the student's waist and shoulders.
  PERFORMANCE CRITERIA:
  Dominant hand grips bat above nondominant hand. Nondominant side of body faces the tossed (feet parallel). Hip and spine rotation. Weight is transferred by stepping with front foot.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Object control skill- stationary bounce | Nine months
  EQUIPMENT/CONDITIONS: An 8-10-inch playground ball and a flat hard surface. DIRECTIONS: Tell the student to bounce the ball three times using one hand. Make sure the ball is not underinflated. Repeat three separate trials.
  PERFORMANCE CRITERIA:
  Contact ball with one hand at about hip height. Pushes ball with fingers (not a slap). Ball contacts floor in front of (or to the outside of) foot on the side of the hand being used.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Object control skill- catch | Nine months
  * EQUIPMENT/CONDITIONS:** A 6-8-inch sponge ball, 15 feet of clear space, masking tape or other marking device.
  * DIRECTIONS:** Mark off two lines 15 feet apart. The student stands on one line, and the ball is tossed from the other. Toss the ball underhand directly to the student with a slight arc, saying "catch it with your hands." Only count tosses between the student's shoulders and waist.
  **PERFORMANCE CRITERIA:**
  1. Preparation phase with elbows flexed and hands in front of the body.
  2. Arms extend in preparation for ball contact.
  3. Ball caught and controlled by hands only.
  4. Elbows bend to absorb force.
  **EXPERT SCORING:**
  1. Require three trials.
  2. Observe and focus on performance criteria.
  3. Score "1" for correct performance on two out of three trials, otherwise score "0."
Test of gross motor development (tgmd-2): Object control skill- kick | Nine months
  EQUIPMENT/CONDITIONS: An 8-10-inch plastic or slightly deflated playground ball, 30 feet of clear space, masking tape or other marking device.
  DIRECTIONS: Mark off two lines-one 30 feet away from a wall and another 20 feet from the wall. Place the ball on the line nearest the wall and have the student stand on the other line. Instruct the student to kick the ball "hard" toward the wall.
  PERFORMANCE CRITERIA:
  Rapid continuous approach to the ball. Trunk inclined backward during ball contact. Forward swing of the arm opposite kicking leg. Follow-through by hopping on non-kicking foot.
  EXPERT SCORING:
  Require three trials. Observe and focus on performance criteria. Score "1" for correct performance on two out of three trials, otherwise score "0."
Test of gross motor development (tgmd-2): Object control skill- overhand throw | Nine months
  EQUIPMENT/CONDITIONS: A tennis ball, a wall, and 25 feet of clear space. DIRECTIONS: Tell the student to throw the ball "hard" at the wall.
  PERFORMANCE CRITERIA:
  A downward arc of the throwing arm initiates the windup. Rotation of hip and shoulder to a point where the nondominant side faces an imaginary target.
  Weight is transferred by stepping with the foot opposite the throwing hand. Follow-through beyond ball release diagonally cross body toward side opposite throwing arm.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."
Test of gross motor development (tgmd-2): Object control skill- underhand roll | Nine months
  EQUIPMENT/CONDITIONS: A tennis ball or a softball; two cones; tape; and 25 feet of clean space.
  DIRECTIONS:
  Place two cones 4 feet apart against a wall. Instruct the child to roll the ball between the cones with force.
  PERFORMANCE CRITERIA:
  Preferred hand swing, reaching behind the trunk while chest faces cones. Strides forward with foot opposite the preferred hand toward the cones. Bends knees to lower body. Releases ball close to the floor so ball does not bounce more than 4 inches high.
  Expert scoring - the specific steps in scoring all items are listed below:
  1. Require the subject to perform three trials.
  2. Observe the student performing the skill and concentrate on the performance criteria.
  3. Where the student performs a behavioural component two out of three trials correctly, mark a "1" in the appropriate box in the correct assessment column. Where the student does not perform a behavioural component two out of three trials correctly, mark "0."

SECONDARY OUTCOMES:
Sex | Nine months
  The sex of the participants is recorded at the start of the study.
Date of birth | Nine months
  The participant's date of birth is collected in order to calculate his age in years.
Weight | Nine months
  The weight of the participants is analyzed in kilograms.
Height | Nine months
  The height of the subject is determined in meters.
Body Mass Index (BMI) | Nine months
  The participant's BMI is calculated from his height and weight.
Adherence | Nine months
  Adherence to the program is calculated from the record of the percentage of attendance at the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Marinkovic, Study Director — University of Novi Sad, Faculty of Sport and Physical Education
Locations (1):
- Faculty of sport and Physical Education, University of Novi Sad, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radanovic D, Marinkovic D, Macak D, Milic Z, Popovic B, Pantovic M, Madic DM. Effects of Developmental Gymnastics Exercise Program on Preschoolers' Motor Skills: A Randomised Controlled Trial. Children (Basel). 2025 Nov 23;12(12):1590. doi: 10.3390/children12121590. PMID 41462731

DOCUMENTS (2):
  • Study Protocol (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT06315036/Prot_000.pdf
  • Informed Consent Form (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT06315036/ICF_001.pdf